CLINICAL TRIAL: NCT01290848
Title: Take TIME for Your Child's Health: A Health Promotion Campaign Targeting Caregivers of Young Children
Brief Title: A Health Promotion Campaign Targeting Caregivers of Young Children
Acronym: TIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other); Township of Uxbridge (Unknown)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000020942
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Childhood Obesity
Keywords: pediatrics; Health Promotion Campaign; Community events
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Township of Uxbridge (Experimental): The Take TIME for Your Child's Health campaign will target parents and caregivers of children up to 8 years of age.
  Interventions: Behavioral: Take TIME Health Campaign
- Township of Guelph/Ermosa (No Intervention): For a control group the investigators have selected a community that is similar in size, household composition, population density, distance from Toronto and economic status to the Township of Uxbridge.

INTERVENTIONS:
Behavioral: Take TIME Health Campaign — 1. Provision of free, family-based events, at least twice per month, that offer opportunities for physical activity and/or healthy eating in a safe, tobacco-free environment.
  2. Information dissemination, via project web site, media and other formats, on how to achieve a healthier lifestyle with the already hectic family schedules.
  3. Adoption of guidelines by community organizations and the Township of Uxbridge that will reduce tobacco exposure, increase safety and promote physical activity and healthy eating for young children.
  Arms: Township of Uxbridge

SUMMARY:
This project will evaluate the effectiveness of the Take TIME health promotion campaign. The Take TIME (Tobacco free, Injury free, Moving daily, Eating healthy) campaign will target parents and caregivers of children up to 8 years of age.

The study will help answer the following research questions

1. Are community organizations able and willing to deliver a health-promotion campaign targeting young children?
2. What impact does the Take TIME campaign have on the readiness of the community to support healthy childhoods?
3. What impact does the Take TIME campaign have on awareness and achievement of healthier lifestyles for young children?
4. Can health promotion initiatives be "institutionalized" within the Municipality and community organizations so that the campaign will continue beyond the study period?
5. Are changes in awareness and/or behaviour related to exposure to the Take TIME campaign?

DETAILED DESCRIPTION:
The Take TIME initiative will be developed and delivered in conjunction with the Township of Uxbridge and the Heart and Stroke Foundation of Ontario. The Durham Region Health Department, the Ministry of Health Promotion and Sport, and 35 schools and community organizations have also agreed to collaborate on project activities. The health promotion campaign will occur from October 15, 2010 until May 31, 2011. The campaign activities were developed from the input of parents and programme/care providers gathered during the planning phase of this research.

The impact of the Take TIME campaign will be evaluated in two ways. The overall readiness of the community to support healthy childhoods will be evaluated using the Community Readiness Model, which relies on a series of interviews with key individuals in leadership positions. Awareness and current behaviour among community members will be assessed through the completion of telephone surveys of randomly selected households. Each of these evaluations will be completed twice, before and after delivery of the Take TIME campaign. The pre-campaign evaluations will be completed in September 2010. The post-campaign evaluations, using the same procedures, will be completed in June 2011.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) or caregiver(s) of young children (8 years of age and younger) will be eligible for the pre- and post- intervention telephone surveys.
* Intervention activities will target parents and caregivers of young children and children 8 years of age and younger, although the events, information and policies may also influence other residents of the community.

Exclusion Criteria:

* Children and adults who are not parents or caregivers for young children 8 years of age or younger are not eligible to complete the random telephone survey.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1374 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Awareness and current behaviour | Baseline
  Household Survey: Randomly selected households will be contacted by telephone to complete the survey questions. The questions address the four key themes of the Take TIME campaign: physical activity, healthy eating, and reducing exposure to injury and tobacco. For each theme, a series of questions are used to assess knowledge, awareness and family behaviour
Awareness and current behaviour | Post-Intervention (9 months)
  Household Survey: Randomly selected households will be contacted by telephone to complete the survey questions. The questions address the four key themes of the Take TIME campaign: physical activity, healthy eating, and reducing exposure to injury and tobacco. For each theme, a series of questions are used to assess knowledge, awareness and family behaviour

SECONDARY OUTCOMES:
Readiness of the community to support healthy childhoods | Baseline, Post-Intervention (9 months)
  A Community Readiness Score will be calculated according to the methods of Findholt for each key stakeholder interview completed. Pre- and post-campaign scores will be compared to determine changes in Community Readiness over the timeframe of the Take TIME for Your Child's Health campaign.
  This second analysis will seek to obtain descriptive information on community strengths and barriers that might impact the success of the Take TIME intervention, and identify similarities and differences between the perspectives of the leader participants.

CONTACTS AND LOCATIONS:
Overall Officials: Brian McCrindle, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Township of Uxbridge, Uxbridge, Ontario